CLINICAL TRIAL: NCT05744921
Title: An Open-Label Extension Study to Evaluate the Long-Term Safety, Tolerability, and Efficacy of Pozelimab and Cemdisiran Combination Therapy in Patients With Paroxysmal Nocturnal Hemoglobinuria
Brief Title: A Study in Adult Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH) to Evaluate How Safe Long-term Treatment With Pozelimab + Cemdisiran Combination Therapy is and How Well it Works
Acronym: ACCESS-EXT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R3918-PNH-2050; 2021-004931-10 (EudraCT Number); 2023-510336-36-00 (EU CTIS Number)
Record Dates: First submitted 2023-02-06; First posted 2023-02-27 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: PNH
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PNH Transition Patients (Experimental): Patients with PNH who completed treatment/ protocol requirements (as applicable) in the parent study (R3918-PNH-2021 [NCT05133531])
  Interventions: Drug: Pozelimab; Drug: Cemdisiran
- C5 Polymorphism Patients (Experimental): Patients who have not been treated in either parent study but who have a documented complement component 5 (C5) variation rendering them refractory to eculizumab/ravulizumab. Note: Loading dose of pozelimab administered IV on Day 1.
  Interventions: Drug: Pozelimab; Drug: Cemdisiran

INTERVENTIONS:
Drug: Pozelimab — Administered per the protocol
  Other Names: REGN3918
Drug: Cemdisiran — Administered per the protocol
  Other Names: ALN-CC5

SUMMARY:
This study is researching an experimental treatment combination with two experimental drugs called pozelimab and cemdisiran. The study is focused on people with paroxysmal nocturnal hemoglobinuria (PNH). The aim of this study is to see how safe and effective the pozelimab + cemdisiran combination is for people with PNH in the long term. The pozelimab + cemdisiran combination may be referred to as "study drugs" in this section.

This study is looking at several other research questions, including:

* How effective is the pozelimab + cemdisiran combination?
* What side effects may happen from taking the study drugs?
* How much of each study drug is in the blood at different times?
* Whether the body makes antibodies against the study drugs (which could make the drugs less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

Patients Entering from the Parent Study

1. Patients with PNH who have completed, without permanent discontinuation, study treatment in the parent study (R3918-PNH-2021[NCT05133531]), including the post-Open-label treatment period (OLTP) transition period, if applicable.
2. Willing and able to comply with clinic visits and study-related procedures, including meningococcal vaccinations required per protocol.

Patients Entering with C5 polymorphism

1. Patients with PNH who have a documented C5 polymorphism rendering them refractory to eculizumab or ravulizumab (eg, p.Arg885His, p.Arg885Cys), as described in the protocol
2. Diagnosis of PNH confirmed by high-sensitivity flow cytometry testing with PNH granulocytes or monocytes
3. Active disease, as defined by the presence of 1 or more PNH-related sign or symptom as described in the protocol
4. LDH level ≥2 × upper limit of normal (ULN) at the screening visit
5. Willing and able to comply with clinic visits and study-related procedures, including meningococcal vaccinations required per protocol

Key Exclusion Criteria:

Patients Entering from the Parent Study

1. Significant protocol deviation(s) in the parent study based on the investigator's judgment and to the extent that these would (if continued) impact the study objectives and/or safety of the patient
2. Any new condition or worsening of an existing condition which, in the opinion of the investigator, would make the patient unsuitable for enrollment or could interfere with the patient participating in or completing the study

Patients Entering with C5 polymorphism

1. Prior treatment with complement inhibitors within 5 half-lives of the respective agent prior to screening, except for prior eculizumab or ravulizumab which are not exclusionary
2. Receipt of an organ transplant, history of bone marrow transplantation or other hematologic transplant
3. Not meeting meningococcal vaccination requirements and, at a minimum, documentation of quadrivalent meningococcal vaccination within 5 years prior to enrollment and serotype B vaccine within 3 years prior to enrollment as described in the protocol
4. Positive hepatitis B surface antigen or hepatitis C virus Ribonucleic acid (RNA) during screening
5. Patients with known HIV with history of opportunistic infections in the last 1 year as described in the protocol
6. Known hereditary complement deficiency
7. Documented history of active, uncontrolled, ongoing systemic autoimmune diseases
8. Documented history of liver cirrhosis or patients with liver disease with evidence of current impaired liver function or patients with elevations in Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) (unrelated to PNH or its complications) as described in the protocol

Note: Other protocol-defined Inclusion/ Exclusion Criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2029-02-26 (Estimated); Study Completion 2029-02-26 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent serious adverse events (SAEs) | Up to week 108
  An SAE is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires in-patient hospitalization or prolongation of existing hospitalization.
  * Results in persistent or significant disability/incapacity
  * Is a congenital anomaly/birth defect.
  * Is an important medical event
Severity of treatment-emergent SAEs | Up to week 108
Incidence of treatment emergent adverse events of special interest (AESIs) | Up to week 108
  An AESI (serious or non-serious) is one of scientific and medical concern specific to the sponsor's product or program, for which ongoing monitoring and rapid communication by the Investigator to the sponsor can be appropriate. Such an event might warrant further investigation in order to characterize and understand it
Severity of treatment emergent AESIs | Up to week 108
Incidence of adverse events (AEs) leading to permanent treatment discontinuation | Up to week 108
  Any untoward medical occurrence in a patient administered a study drug which may or may not have a causal relationship with the study drug.
Severity of adverse events (AEs) leading to permanent treatment discontinuation | Up to week 108
  Any untoward medical occurrence in a patient administered a study drug which may or may not have a causal relationship with the study drug.
Percent change from baseline in lactate dehydrogenase (LDH) | Baseline to week 36

SECONDARY OUTCOMES:
Adequate control of hemolysis (LDH ≤1.5 × ULN) | Post-baseline through week 108
Transfusion avoidance | Post-baseline through week 36
  Not requiring red blood cell (RBC) transfusion as per protocol algorithm based on hemoglobin values
Transfusion avoidance | Post-baseline through week 48
  Not requiring red blood cell (RBC) transfusion as per protocol algorithm based on hemoglobin values
Transfusion avoidance | Post-baseline through week 76
  Not requiring red blood cell (RBC) transfusion as per protocol algorithm based on hemoglobin values
Transfusion avoidance | Post-baseline through week 108
  Not requiring red blood cell (RBC) transfusion as per protocol algorithm based on hemoglobin values
Breakthrough hemolysis (defined as LDH ≥2 × ULN [subsequent to initial achievement of LDH ≤1.5 × ULN] concomitant with signs or symptoms associated with hemolysis) | Post-baseline through week 36
Breakthrough hemolysis (defined as LDH ≥2 × ULN [subsequent to initial achievement of LDH ≤1.5 × ULN] concomitant with signs or symptoms associated with hemolysis) | Post-baseline through week 48
Breakthrough hemolysis (defined as LDH ≥2 × ULN [subsequent to initial achievement of LDH ≤1.5 × ULN] concomitant with signs or symptoms associated with hemolysis) | Post-baseline through week 76
Breakthrough hemolysis (defined as LDH ≥2 × ULN [subsequent to initial achievement of LDH ≤1.5 × ULN] concomitant with signs or symptoms associated with hemolysis) | Post-baseline through week 108
Hemoglobin stabilization | Post-baseline through week 36
  Patients who do not receive an RBC transfusion and have no decrease in hemoglobin level of ≥2 g/dL
Hemoglobin stabilization | Post-baseline through week 48
  Patients who do not receive an RBC transfusion and have no decrease in hemoglobin level of ≥2 g/dL
Hemoglobin stabilization | Post-baseline through week 76
  Patients who do not receive an RBC transfusion and have no decrease in hemoglobin level of ≥2 g/dL
Hemoglobin stabilization | Post-baseline through week 108
  Patients who do not receive an RBC transfusion and have no decrease in hemoglobin level of ≥2 g/dL
Percent change in LDH | From baseline to week 48
Percent change in LDH | From baseline to week 76
Percent change in LDH | From baseline to week 108
Change in fatigue | From baseline to week 36
  Measured by the FACIT-Fatigue scale The FACIT-F is a 13-item, self-reported PRO measure assessing an individual's level of fatigue during their usual daily activities over the past week. This questionnaire is part of the FACIT measurement system, a compilation of questions measuring health-related QoL in patients with cancer and other chronic illnesses. The FACIT-fatigue assesses the level of fatigue using a 5-point Likert scale ranging from 0 (not at all) to 4 (very much). Scores range from 0 to 52, with higher scores indicating greater fatigue.
Change in fatigue | From baseline to week 48
  Measured by the FACIT-Fatigue scale The FACIT-F is a 13-item, self-reported PRO measure assessing an individual's level of fatigue during their usual daily activities over the past week. This questionnaire is part of the FACIT measurement system, a compilation of questions measuring health-related QoL in patients with cancer and other chronic illnesses. The FACIT-fatigue assesses the level of fatigue using a 4-point Likert scale ranging from 0 (not at all) to 4 (very much). Scores range from 0 to 52, with higher scores indicating greater fatigue.
Change in fatigue | From baseline to week 76
  Measured by the FACIT-Fatigue scale The FACIT-F is a 13-item, self-reported PRO measure assessing an individual's level of fatigue during their usual daily activities over the past week. This questionnaire is part of the FACIT measurement system, a compilation of questions measuring health-related QoL in patients with cancer and other chronic illnesses. The FACIT-fatigue assesses the level of fatigue using a 4-point Likert scale ranging from 0 (not at all) to 4 (very much). Scores range from 0 to 52, with higher scores indicating greater fatigue.
Change in fatigue | From baseline to weeks 108
  Measured by the FACIT-Fatigue scale The FACIT-F is a 13-item, self-reported PRO measure assessing an individual's level of fatigue during their usual daily activities over the past week. This questionnaire is part of the FACIT measurement system, a compilation of questions measuring health-related QoL in patients with cancer and other chronic illnesses. The FACIT-fatigue assesses the level of fatigue using a 4-point Likert scale ranging from 0 (not at all) to 4 (very much). Scores range from 0 to 52, with higher scores indicating greater fatigue.
Change in physical function (PF) scores on the EORTC QLQ-C30 | From baseline to week 36
  EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire)
  EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including a global health status/quality of life (GHS/QoL) scale. Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change.
Change in PF scores on the EORTC QLQ-C30 | From baseline to week 48
  EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire)
  EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including a global health status/quality of life (GHS/QoL) scale. Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change.
Change in PF scores on the EORTC QLQ-C30 | From baseline to week 76
  EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire)
  EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including a global health status/quality of life (GHS/QoL) scale. Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change.
Change in PF scores on the EORTC QLQ-C30 | From baseline to week 108
  EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire)
  EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including a global health status/quality of life (GHS/QoL) scale. Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change.
Change in GHS/quality of life (QOL) scale on the EORTC QLQ-C30 | From baseline to week 36
  GHS/QoL (Global Health Status/ Quality of Life)
  Global Health Status/Quality of Life (GHS/Qol) Score (Items 29 and 30) Using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change.
Change in GHS/quality of life (QOL) scale on the EORTC QLQ-C30 | From baseline to week 48
  GHS/QoL (Global Health Status/ Quality of Life)
  Global Health Status/Quality of Life (GHS/Qol) Score (Items 29 and 30) Using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change.
Change in GHS/quality of life (QOL) scale on the EORTC QLQ-C30 | From baseline to week 76
  GHS/QoL (Global Health Status/ Quality of Life)
  Global Health Status/Quality of Life (GHS/Qol) Score (Items 29 and 30) Using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change.
Change in GHS/quality of life (QOL) scale on the EORTC QLQ-C30 | From baseline to week 108
  GHS/QoL (Global Health Status/ Quality of Life)
  Global Health Status/Quality of Life (GHS/Qol) Score (Items 29 and 30) Using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change.
Normalization of LDH | From post-baseline through week 108
Rate of red blood cell (RBC) transfusion | Post-baseline through week 36
  Per protocol algorithm
Rate of RBC transfusion | Post-baseline through week 48
  Per protocol algorithm
Rate of RBC transfusion | Post-baseline through week 76
  Per protocol algorithm
Rate of RBC transfusion | Post-baseline through week 108
  Per protocol algorithm
Number of units of RBC transfusion | Post-baseline through week 36
  Per protocol algorithm
Number of units of RBC transfusion | Post-baseline through week 48
  Per protocol algorithm
Number of units of RBC transfusion | Post-baseline through week 76
  Per protocol algorithm
Number of units of RBC transfusion | Post-baseline through week 108
  Per protocol algorithm
Percentage of days with LDH ≤1.5x upper limit of normal (ULN) | Post-baseline through week 36
Percentage of days with LDH ≤1.5x ULN | Post-baseline through week 48
Percentage of days with LDH ≤1.5x ULN | Post-baseline through week 76
Percentage of days with LDH ≤1.5x ULN | Post-baseline through week 108
Change in hemoglobin levels | From baseline to week 36
Change in hemoglobin levels | From baseline to week 48
Change in hemoglobin levels | From baseline to week 76
Change in hemoglobin levels | From baseline to week 108
Change in total complement hemolytic activity assay (CH50) | Through week 108
Percent change in CH50 | Through week 108
Concentrations of total pozelimab in serum | Through week 108
Concentrations of cemdisiran in plasma | Through week 24
Incidence of treatment-emergent anti-drug antibodies to pozelimab | Through week 108
Incidence of treatment-emergent anti-drug antibodies to cemdisiran | Through week 108
Concentration of total complement component 5 (C5) in plasma | Through week 108
Percent change of concentration of total C5 in plasma | Through week 108

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (41):
- Toronto General Hospital, Toronto, Ontario, Canada
- Hospital Pablo Tobon Uribe, Medellín, Antioquia, Colombia
- Semmelweis University/Semmelweis Egyetem, Budapest, Hungary
- India (4):
  - Amrita Institute of Medical Sciences (AIMS) and Research Centre Aims, Kochi, Kerala
  - K J Somaiya Super Specialty Hospital & Research Centre, Mumbai, Maharashtra
  - Rajiv Gandhi Cancer Institute & Research Center (RGCIRC) - Rohini Campus, New Delhi, National Capital Territory of Delhi
  - Bhagwan Mahaveer Cancer Hospital and Research Centre (BMCHRC), Jaipur
- Italy (2):
  - Aou Careggi, Florence, Firenze
  - SC Hematology, AOU Città della Salute e della Scienza di Torino, Torino
- University of Tsukuba Hospital, Tsukuba, Ibaraki, Japan
- Jordan University Hospital (JUH), Amman, Jordan
- Malaysia (3):
  - Hospital Tg Ampuan Afzan, Kuantan, Pahang
  - Hospital Queen Elizabeth, Kota Kinabalu, Sabah
  - Hospital Ampang, Ampang, Selangor
- Clinica San Felipe, Lima, Peru
- St Lukes Medical Center, Quezon City, National Capital Region, Philippines
- Poland (3):
  - IN-VIVO Sp. z o.o., Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - University Clinical Center Medical University of Gdansk, Gdansk, Pomeranian Voivodeship
  - Szpital Uniwersytecki Nr2 Bydgoszcz, Bydgoszcz
- Prof Dr Ion Chiricuta Cancer Institute, Cluj-Napoca, Cluj, Romania
- National University Hospital, Singapore, Singapore
- South Korea (7):
  - St. Vincent Hospital, Suwon, Gyeonggi-do
  - Ajou University Medical Center, Suwon, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon, Namdong-Gu
  - Pusan National University Hospital, Busan
  - Severance Hospital Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
- Spain (2):
  - Hospital Universitario Basurto, Bilbao, Vizcaya
  - Hospital Clinic de Barcelona, Barcelona
- Taiwan (5):
  - China Medical University Hospital, Taichung, Central Taiwan
  - Chang Gung Memorial Hospital - Linkou Branch, Taoyuan District, Hunan Province
  - Hualien Tzu Chi Hospital, Hualien City
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
- Thailand (4):
  - Prince Of Songkla Hospital, Prince Of Songkhla University, Hat Yai, Changwat Songkhla
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Chiang Mai University, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
- Ege University Faculty of Medicine, Bornova, İzmir, Turkey (Türkiye)
- Leeds Teaching Hospitals NHS Trust - St. James Institute of Oncology, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry),
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/